CLINICAL TRIAL: NCT06647537
Title: Frequency of Neonatal Hyperglycemia at Assuit University Children Hospital
Brief Title: Frequency of Neonatal Hyperglycemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Rashad abdeltawab, doctor, Assiut University
Other Study IDs: Neonatal hyperglycemia
Record Dates: First submitted 2024-09-24; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Hyperglycemia
Keywords: Neonatal hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detection of prevalence of neonatal hyperglycemia and assessment of risk factors, clinical characteristics and possible complications of neonatal hyperglycemia.

DETAILED DESCRIPTION:
Hyperglycemia has become an important risk factor for mortality and morbidity in the neonatal period, especially with increased survival rates of very low birth weight neonates.

Neonatal hyperglycemia is usually defined as serum glucose greater than 150 mg/dl (8.3 mmol/L) or whole blood glucose greater than 125 mg/dl (6.9 mmol/L) irrespective of gestational or postmenstrual age. Usually, the safe target for a neonate's serum glucose level is 70 to 150 mg/dl. The cut off for safe target is based on the renal glucose threshold of preterm neonates.

Hyperglycemia is more common in preterm infants than term infants as it occurs in one-third of preterm and small gestational age (SGA) infants and is generally noted during the first week of life. Usually, the acute hyperglycemia resolves over two to three days in most neonates but can last up to ten days. Hyperglycemia is less common than hypoglycemia among neonates but is associated with increased mortality and morbidity among neonates. Neonatal hyperglycemia is inversely related to birth weight and gestational age.

Glucose is an essential source of energy for the fetus and neonate. The brain growth of the fetus exclusively depends upon glucose. In the early postnatal period, glucose homeostasis occurs via glycogenolysis and gluconeogenesis. The critical regulatory mechanisms of glucose homeostasis are sluggish in the initial days, particularly among preterm neonates. The mechanisms of neonatal hyperglycemia are multifactorial. The risk of hyperglycemia increases with the severity of the accompanying illness. The most common cause is high exogenous glucose infusion rates (GIR) in preterm infants who are already at risk for hyperglycemia due to the following reasons,

* decreased ability to suppress endogenous glucose production,
* decreased insulin response to glucose, and
* limited glycogen and fat stores. Hyperglycemia in the neonatal period develops as a result of other multiple risk factors including.

Intrauterine growth restriction, increased stress hormones like epinephrine and norepinephrine inhibit both insulin secretion and action, causes related to enteral feeding as delay in the initiation of enteral feeding causes decreased incretin secretion, which in turn causes hyperglycemia. and the hyperosmolar formula may lead to transient glucose intolerance in the baby. , causes related to Total parenteral nutrition (TPN) as delay in supplementing parenteral amino acids in TPN delays the release of insulin-like growth factor-1, which delays the development of beta cells in the pancreas and develops hyperglycemia and a high intravenous lipid infusion rate causes an increase in free fatty acids (FFA), which decrease glucose oxidation competitively by providing additional carbon substrates for oxidative metabolism. FFA and glycerol promote gluconeogenesis, sepsis, iatrogenic as error in the glucose infusion rate (GIR) calculation in the intravenous (IV) fluid, transient neonatal diabetes mellitus and permanent diabetes mellitus, drugs as maternal medications as maternal Diazoxide may cause hyperglycemia, hypotension, and tachycardia in neonates, antenatal steroids, neonatal medications as dopamine, dobutamine, epinephrine infusions, caffeine, theophylline, Phenytoin and Corticosteroids.

Neonatal diabetes can be of three different types.

1. The transient form accounts for more than 50%. It is usually associated with mutations of sulfonylurea receptors. Transient neonatal diabetes manifests soon after birth and remits spontaneously in 6 months.
2. Permanent neonatal diabetes needs lifelong management. Mutations in the genes encoding the subunit of the ATP-sensitive potassium channel is the most common cause.
3. Syndromic Neonatal diabetes is usually associated with syndromes like Wolfram syndrome, IPEX syndrome (immune dysregulation polyendocrinopathy X linked syndrome).

The severity of impact increases with prolonged hyperglycemia as intracranial hemorrhage by causing hyperosmolarity with osmotic shifts, dehydration due to osmotic diuresis, electrolyte imbalance occurs due to osmotic diuresis. Glycosuria also increases sodium excretion, NEC , retinopathy of prematurity , bronchopulmonary disease, Impaired immunity and increased risk of sepsis, poor wound healing and adverse neurodevelopmental outcome.

In general, Neonatal hyperglycemia is associated with a clinical condition rather than a specific disorder of glucose metabolism. Neonatal hyperglycemia can be a sign of an underlying illness.

In preterm and very-low-birth-weight (VLBW) infants, i.e., infants with birth weight less than 1500 grams, a consistent blood glucose level of more than 200 mg/dL is a cause for concern. A blood glucose level measured as >200 mg/dL with a 4-hour interval and glucosuria of +2 or more necessitates treatment. Currently, hyperglycemia treatment in the absence of an increase in osmolarity and osmotic diuresis is not supported.

1. The first step in evaluating neonatal hyperglycemia is to assess the GIR. GIR = IV infusion rate (mL/kg/day) x Dextrose concentration (%) / 144 The GIR is lowered by reducing IV dextrose concentration or the infusion rate. GIR can be decreased by 1 to 2 mg/kg/min every 2 hours, with frequent glucose monitoring until the GIR reaches 4 mg/kg/min.
2. In case of persistent hyperglycemia, underlying causes such as sepsis, stress, medications need to be explored and treated accordingly.
3. Role of Insulin

   * Hyperglycemia persisting at low GIR (4 mg/kg/min) may indicate relative insulin deficiency or insulin resistance.
   * The role of insulin therapy in treating hyperglycemia in neonates is controversial. Consider insulin if blood glucose level is more than 250 mg/dl, and if urine glucose is more than 2+ in two separate samples obtained four hours apart.
   * It is crucial to monitor serum glucose levels every 1 hour when the infant is on insulin. Measure the blood glucose level half an hour after each change in insulin infusion
4. Any electrolyte imbalance due to osmotic diuresis should be corrected. Sodium and potassium imbalance is very common.

Hyperglycemia needs to be prevented in all neonates, particularly among preterm infants, due to associated complications such as the increased risk for infection, impaired immunity, poor wound healing, increased morbidity, and mortality. The following preventive measures help in the practice to prevent hyperglycemia.

1. Early initiation of enteral feedings
2. Early supplementation of amino acids in TPN, leading to an increase in insulin secretion that prevents hyperglycemia.
3. Targeting optimal and physiologic GIR in TPN as per the glucose monitoring
4. Limiting IV lipid infusions during hyperglycemia
5. A more direct and immediate approach is to decrease the catecholamine infusions as tolerated.
6. Discontinuing catecholamine infusions and glucocorticoid treatments as soon as the infant;s condition has improved.

ELIGIBILITY:
Inclusion Criteria:

* all neonates from day 0 to 28 days old admitted in NICU.

Exclusion Criteria:

* > 28 days old

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: - all neonates from day 0 to 28 days old admitted in NICU.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1-Detection of prevalence of neonatal hyperglycemia by estimating RBG level in serum 2-Assessment of risk factors, clinical characteristics and possible complications of neonatal hyperglycemia. | 1_11_2024
  assesment how many children diagnosed with neonatal hyperglycemia . what are risk factors those cause this problem . what are the manifestationsof neonatal hyperglycemia and possible complications of neonatal hyperglycemia
1-Detection of prevalence of neonatal hyperglycemia by estimating RBG level in serum 2-Assessment of risk factors, clinical characteristics and possible complications of neonatal hyperglycemia. | 1-11-2024
  assesment how many children diagnosed with neonatal hyperglycemia . what are risk factors those cause this problem . what are the manifestationsof neonatal hyperglycemia and possible complications of neonatal hyperglycemia

REFERENCES:
- [Background] Kao LS, Morris BH, Lally KP, Stewart CD, Huseby V, Kennedy KA. Hyperglycemia and morbidity and mortality in extremely low birth weight infants. J Perinatol. 2006 Dec;26(12):730-6. doi: 10.1038/sj.jp.7211593. Epub 2006 Aug 24. PMID 16929344
- [Background] Sunehag AL, Haymond MW. Glucose extremes in newborn infants. Clin Perinatol. 2002 Jun;29(2):245-60. doi: 10.1016/s0095-5108(02)00006-4. No abstract available. PMID 12168240
- [Background] Mitanchez D. Glucose regulation in preterm newborn infants. Horm Res. 2007;68(6):265-71. doi: 10.1159/000104174. Epub 2007 Jun 20. PMID 17587854